CLINICAL TRIAL: NCT02381652
Title: An Open-Label, Follow-On Study to Cingal 13-01 to Evaluate the Safety of a Repeat Injection of Cross-Linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide to Provide Symptomatic Relief of Osteoarthritis of the Knee
Brief Title: Repeat Injection of Cingal® for Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cingal 13-02
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Intra-articular Injection; Hyaluronic Acid; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid; triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: All subjects enrolled into the Cingal 3-02 follow-on study received an intra-articular injection of Cingal. The three 'arms' of the study were for subjects who received a Cingal, Monovisc, or saline initial injection in the Cingal 13-01 study.
Masking Description: Cingal 13-02 was an open label follow-up study. The participants, investigators and outcomes assessors were blinded to the specific study injection subjects had previously received in Cingal 13-01.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cingal/Cingal (Experimental): Subjects who had received an injection of Cingal in the 13-01 study will receive a single 4 milliliter (mL) intra-articular injection of Cingal (88 milligrams Hyaluronic Acid plus 18 milligramsTriamcinolone Hexacetonide) in the index knee in the 13-02 study.
  Interventions: Combination Product: Cingal
- Cingal/Monovisc (Experimental): Subjects who had received an injection of Monovisc in the 13-01 study will receive a single 4 milliliter (mL) intra-articular injection of Cingal (88 milligrams Hyaluronic Acid plus 18 milligramsTriamcinolone Hexacetonide) in the index knee in the 13-02 study.
  Interventions: Combination Product: Cingal
- Cingal/Saline (Experimental): Subjects who had received an injection of Saline in the 13-01 study will receive a single 4 milliliter (mL) intra-articular injection of Cingal (88 milligrams Hyaluronic Acid plus 18 milligramsTriamcinolone Hexacetonide) in the index knee in the 13-02 study.
  Interventions: Combination Product: Cingal

INTERVENTIONS:
Combination Product: Cingal — Injection into the knee
  Other Names: Hyaluronic Acid with Triamcinolone Hexacetonide
  Arms: Cingal/Cingal
Combination Product: Cingal — Injection into the knee
  Other Names: Hyaluronic Acid with Triamcinolone Hexacetonide
  Arms: Cingal/Monovisc
Combination Product: Cingal — Injection into the knee
  Other Names: Hyaluronic Acid with Triamcinolone Hexacetonide
  Arms: Cingal/Saline

SUMMARY:
The objective of this study is to evaluate the safety of an injection of Cingal® in subjects with Osteoarthritis (OA) of the knee who participated in Cingal 13-01, and who received either a Cingal, Monovisc, or saline injection in the 13-01 study. The safety evaluation will be done by a through examination of the incidence of adverse events and physical examination of the knee.

DETAILED DESCRIPTION:
The Cingal 13-02 study is a follow-on study to the recently completed clinical trial Cingal 13-01 [NCT01891396]. Cingal 13-01 was a multi-center, randomized, double-blind, Phase III study that enrolled 368 subjects at up to 20 sites in Canada and Europe. The Cingal 13-01 study objective was to assess the safety and effectiveness of a single injection of Cingal® for relief of joint pain and symptoms in patients with osteoarthritis (OA) of the knee. The study had three arms: the Cingal® investigational arm, an active comparator arm (Monovisc®) and a control arm (saline). Cingal 13-02 is designed to evaluate the safety of an open-label injection of Cingal® in subjects who received a study injection in the Cingal 13-01 trial. Sites that enrolled 5 or more subjects in the Cingal 13-01 study were eligible to participate in the Cingal 13-02 study. All subjects at these sites who met enrollment criteria had the option to participate in the follow-on study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject completed Cingal 13-01 and is interested in participating in the follow-on study
2. Subject must be willing to abstain from other intra-articular or surgical treatments of the index knee for the duration of the study
3. Subject is willing to discontinue all analgesics except acetaminophen/paracetamol for the duration of the study
4. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least twenty-four hours prior to the injection and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol
5. Subject is able to understand and comply with the requirements of the study and voluntarily provides consent

Exclusion Criteria:

1. Subject received an intra-articular injection or underwent a surgical procedure of the index knee since the study injection in Cingal 13-01
2. Subject is taking medication at the time of consent which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment and opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
3. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index knee only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index knee is allowed.
4. Subject has a contraindication to IA injections, aspiration of the index knee, corticosteroids, hyaluronan, or acetaminophen/paracetamol.
5. Subject is pregnant or breastfeeding or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
6. Subject participated in a research study other than Cingal 13-01 within 60 days of consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, PhD, DSc, Principal Investigator — Semmelweis University, Head of Department of Traumatology; Piotr Lukasik, MD, PhD, Principal Investigator — NZOZ Medi-Spatz
Locations (10):
- Medical Plus s.r.o., Uherské Hradiště, Czechia
- Hungary (6):
  - Belvaros-Lipotvaros, Orthopedic Outpatient Clinic, Budapest
  - Semmelweis University, Department of Orthopaedics, Budapest
  - Uzsoki Hospital, Department of Traumatology, Budapest
  - Jutrix Healthcare Services Ltd., Kecskemét
  - Medidea Bt., Kiskunfélegyháza
  - G&V Pharma-Med Bt., Makó
- Poland (3):
  - NZOZ Medi-Spatz, Gliwice
  - ARTIMED Niepubliczny Zaklad Opieki Zdrowotnej w Kielcach, Kielce
  - CenterMed Krakow Sp. z o.o., Krakow

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited into Cingal 13-02 in February 2015. Sites that enrolled 5 or more subjects in the Cingal 13-01 study were eligible to participate in the Cingal 13-02 study. All subjects at these sites who met enrollment criteria had the option to participate in the follow-on study.
Pre-assignment Details: All enrolled subjects were treated with Cingal in the study. There were no exclusions.
Period: Overall Study
Arm/Group | Cingal/Cingal | Cingal/Monovisc | Cingal/Saline
Started (Safety Population and Intent to Treat Population consisted of all enrolled subjects) | 94 (Cingal injection in 13-01 study; receiving a 2nd Cingal injection in 13-02) | 98 (Monovisc injection in 13-01 study; receiving a Cingal injection in 13-02) | 50 (Saline injection in 13-01 study; receiving a Cingal injection in 13-02)
Completed | 94 | 98 | 49
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population is the Safety Population and consists of all 242 enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Cingal/Cingal | Cingal/Monovisc | Cingal/Saline | Total
Number analyzed (Participants) | 94 | 98 | 50 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (8.2) | 60.2 (8.4) | 60.5 (8.8) | 59.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 68 | 38 | 161
  Male | 39 | 30 | 12 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 94 | 98 | 50 | 242
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events: Cingal 13-02 vs. Cingal 13-01
Description: The primary outcome measure will compare safety results (all adverse events, whether related to the study injection or not) for Cingal 13-01 and Cingal 13-02.
Time Frame: Baseline through 6 weeks post-injection
Population: NOTE: All subjects enrolled in Cingal 13-02 were initially also enrolled in Cingal 13-01 [NCT01891396]. Detail on adverse events that occurred in Cingal 13-01 [NCT01891396] may be found in the summary for that study on clinicaltrials.gov.
Measure: Number; unit: Adverse events
Groups:
- Cingal 13-02 Adverse Events: All adverse events that occurred in Cingal 13-02 for 6 weeks post-injection, regardless if considered related to the study injection or not.
Arm/Group | Cingal 13-02 Adverse Events
Number analyzed (Participants) | 242
Adverse events | 73
Statistical Analysis 1: Comparison: Cingal 13-02 Adverse Events; Test type: Other — Statistical test to see if there is a difference; p = 0.3108, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected in Cingal 13-02 within the first six weeks after injection.
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions. The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Cingal/Cingal | Cingal/Monovisc | Cingal/Saline
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/98 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/98 | 0/50
Other Adverse Events (participants affected / at risk) | 17/94 | 20/98 | 13/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal/Cingal (N=94) | Cingal/Monovisc (N=98) | Cingal/Saline (N=50)
Meniscus injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Subject 18-044 received an injection of Cingal® in the left knee, and 18 days later the subject was hospitalized for a meniscus lesion of the right (non-index) knee. The subject had an arthroscopy and the event resolved without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cingal/Cingal (N=94) | Cingal/Monovisc (N=98) | Cingal/Saline (N=50)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 5 — Generalized joint pain
Nasopharyngitis (Infections and infestations) | 4 | 4 | 1 — Common cold
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 — Swollen knee
Headache (Nervous system disorders) | 1 | 3 | 2 — Headache
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 — Limitation of joint movement
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 — Backache
Injection site pain (General disorders) | 0 | 2 | 1 — Pain at injection site

LIMITATIONS AND CAVEATS:
Cingal 13-02 is a follow-on safety trial to Cingal 13-01 and collected safety data only from an open-label injection of Cingal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No